CLINICAL TRIAL: NCT06740955
Title: A Randomized, Open, Controlled, Multi-center Clinical Trial of Hypofractionated Postoperative Radiotherapy for Adult Glioblastoma
Brief Title: Hypofractionated Radiotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HR-3
Record Dates: First submitted 2024-12-15; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-08

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Experimental group (Experimental): subjects randomly assigned to the experimental group were required to start treatment within 7 working days. The experimental group received hypofractionated radiotherapy with a total dose of 52.5Gy, 3.5 Gy/ fraction, 15 fractions, 5 fractions per week, and temozolomide was given for 21 days. Sequential temozolomide chemotherapy was started 4 weeks after the end of chemoradiotherapy. Sequential chemotherapy was given 5 days before each 28-day cycle.
  Interventions: Radiation: hypofractionated postoperative radiotherapy
- Control group (Other): subjects randomly assigned to the experimental group were treated within 7 working days. The control group received conventional fractionated radiotherapy with a dose of 60Gy, 2Gy per fraction, 30 fractions, 5 fractions per week, and temozolomide was given for a total of 42 days. Sequential temozolomide chemotherapy was started 4 weeks after the end of chemoradiotherapy. Sequential chemotherapy was given 5 days before each 28-day cycle.
  Interventions: Radiation: Conventionally fractionated postoperative radiotherapy

INTERVENTIONS:
Radiation: hypofractionated postoperative radiotherapy — hypofractionated radiotherapy with a total dose of 52.5Gy, 3.5 Gy/ fraction, 15 fractions, 5 fractions per week,
  Arms: Experimental group
Radiation: Conventionally fractionated postoperative radiotherapy — Conventionally fractionated radiotherapy with a total dose of 60 Gy, 2 Gy/ fraction, 30 fractions, 5 fractions per week,
  Arms: Control group

SUMMARY:
This study was a multicenter, open-label, randomized, controlled, phase Ⅲ clinical trial to evaluate the efficacy and safety of hypofractionated concurrent radiotherapy followed by sequential temozolomide after surgery in patients with newly diagnosed glioblastoma.

A total of 420 subjects were enrolled in this study, randomized 1:1. According to the changes in overall survival time after postoperative concurrent chemoradiotherapy with different radiation doses, the stratification factors included the extent of surgical resection (total resection vs subtotal resection); The time of postoperative concurrent chemoradiotherapy (less than 28 days or more than 28 days); MGMT promoter methylation expression (positive or negative).

The study design was as follows: Participants were required to undergo a screening period within 14 days before randomization to determine eligibility. Subjects who met the inclusion criteria were randomly divided into two groups at a 1:1 ratio: trial group, hypofractionated concurrent chemoradiotherapy followed by at least 6 cycles of adjuvant temozolomide; The control group was treated with the existing standardized treatment (standard dose of concurrent chemoradiotherapy and at least 6 cycles of temozolomide adjuvant chemotherapy).

Experimental group: subjects randomly assigned to the experimental group were required to start treatment within 7 working days. The experimental group received hypofractionated radiotherapy with a total dose of 52.5Gy, 3.5 Gy/ fraction, 15 fractions, 5 fractions per week, and temozolomide was given for 21 days. Sequential temozolomide chemotherapy was started 4 weeks after the end of chemoradiotherapy. Sequential chemotherapy was given 5 days before each 28-day cycle. During the study period, the experimental group was required to complete the vital signs, physical examination, laboratory examination and other examinations within the specified period. After randomization, the experimental group underwent radiologic response assessments (or as deemed necessary by the investigator based on clinical symptoms) and QOLs at the end of radiotherapy, 3-4 weeks after the end of radiotherapy, and every 12 weeks (±7 days). Radiologic response assessments required plain and contrast-enhanced magnetic resonance imaging. If there were residual lesions after surgery, measurable lesions were evaluated according to RANO standard case criteria.

Control group: subjects randomly assigned to the experimental group were treated within 7 working days. The control group received conventional fractionated radiotherapy with a dose of 60Gy, 2Gy per fraction, 30 fractions, 5 fractions per week, and temozolomide was given for a total of 42 days. Sequential temozolomide chemotherapy was started 4 weeks after the end of chemoradiotherapy. Sequential chemotherapy was given 5 days before each 28-day cycle. During the study period, the experimental group was required to complete the vital signs, physical examination, laboratory examination and other examinations within the specified period. After randomization, the experimental group underwent radiologic response assessments (or as deemed necessary by the investigator based on clinical symptoms) and QOLs at the end of radiotherapy, 3-4 weeks after the end of radiotherapy, and every 12 weeks (±7 days). Radiologic response assessments required plain and contrast-enhanced magnetic resonance imaging. Measurable lesions assessed according to RANO criteria were required if residual lesions were present after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed glioblastoma confirmed by histopathology or molecular pathology;
2. Complete or partial tumor resection or biopsy via neurosurgery;
3. The age of signing the informed consent form was 18-70 years old, male or female; (4) KPS score ≥60; (5) expected survival time ≥6 months;

6. Radiotherapy should be started within 6 weeks after surgery; 7. Vital organ function meets the following requirements (excluding the use of any blood components and cell growth factors within 14 days) : Normal bone marrow reserve: white blood cell (WBC) ≥3.0×109/L, neutrophil count (NEUT) ≥1.5×109/L, platelet count (PLT) ≥80×109/L, hemoglobin (Hb) ≥90 g/L Normal renal function or serum creatinine (SCr) ≤ 1.5 times the upper limit of normal (ULN) or creatinine clearance ≥50 ml/ minute (Cockcroft-Gault equation) Normal liver function or total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN) Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≤ 2.5 times the upper limit of normal (ULN); 8. Able and willing to follow the study and follow-up procedures; 9. Men and women of childbearing potential must agree to use adequate contraception throughout the study and for 6 months after the end of treatment. Female subjects of childbearing potential were required to have a negative blood pregnancy test within 72 hours before the first dose.

10. The subjects voluntarily participated in this clinical study and signed the informed consent form. The compliance was good and the subjects could cooperate with the follow-up.

Exclusion Criteria:

1. Received any previous systemic antitumor therapy against the target lesion;
2. Prior radiation therapy to the head;
3. Had a history of low-grade glioma and the current tumor transitioned to glioblastoma;
4. The patient had glioma in other parts in the past, and now had metastasis, and the metastatic site was glioblastoma.
5. Subjects were unable to undergo MRI examination or unable to undergo enhanced MRI examination.
6. Patients who received bevacizumab or iodine internal radiation within one month before enrollment;
7. Participants who participated in other clinical trials within 1 month before enrollment;
8. Subjects with severe trauma or severe infection within 1 month before enrollment, including but not limited to infectious complications requiring hospitalization, bacteremia, severe pneumonia, etc.
9. Severe cardiovascular disease: grade Ⅱ or above myocardial ischemia or myocardial infarction, uncontrolled arrhythmia (QTc interval ≥ 450 ms in men and ≥ 470 ms in women); Patients with grade ⅲ-ⅳ cardiac dysfunction (according to the New York Heart Association NYHA classification, see Appendix 3) or left ventricular ejection fraction (LVEF) less than 50% on echocardiography;
10. Subjects underwent major surgery (excluding glioma surgery) within 4 weeks before enrollment;
11. The subjects had a history of psychotropic drug abuse or drug use;
12. Patients with other malignant tumors within 5 years before enrollment (if cured) were excluded;
13. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active hepatitis B (HBV DNA≥500 IU/ml), hepatitis C (hepatitis C antibody positive and HCV-RNA higher than the detection limit of the analytical method) or co-infection with hepatitis B and C;
14. Subjects were allergic to temozolomide or could not receive temozolomide treatment for other reasons;
15. The results of blood pregnancy test of female subjects during non-lactation period and within 7 days before the first study treatment were positive. The subject (male or female) declined to commit to using at least one acceptable contraceptive method (i.e., using an intrauterine device (IUD), condom, any form of hormonal contraceptive, or abstinence, etc.) for the entire duration of the study and for 3 months after the last study treatment;
16. Other conditions that increase the risk associated with participating in the study or the study drug and, in the investigator's judgment, may make the subject ineligible for the study;
17. The investigator determined that he was not fit to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 18 months
  It was defined as the time between the start of the randomization date and the death of the subject due to various causes.

SECONDARY OUTCOMES:
Progression-free survival | 12 months
  The experimental and control groups were defined as the time from randomization to tumor progression (according to RANO criteria) or death from any cause, whichever occurred first.
Time to disease progression | 12 months
  Interval between the date of randomization and the occurrence of radiographic progression according to RANO criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panet-Raymond V, Souhami L, Roberge D, Kavan P, Shakibnia L, Muanza T, Lambert C, Leblanc R, Del Maestro R, Guiot MC, Shenouda G. Accelerated hypofractionated intensity-modulated radiotherapy with concurrent and adjuvant temozolomide for patients with glioblastoma multiforme: a safety and efficacy analysis. Int J Radiat Oncol Biol Phys. 2009 Feb 1;73(2):473-8. doi: 10.1016/j.ijrobp.2008.04.030. Epub 2008 Jun 12. PMID 18554821
- [Background] Sultanem K, Patrocinio H, Lambert C, Corns R, Leblanc R, Parker W, Shenouda G, Souhami L. The use of hypofractionated intensity-modulated irradiation in the treatment of glioblastoma multiforme: preliminary results of a prospective trial. Int J Radiat Oncol Biol Phys. 2004 Jan 1;58(1):247-52. doi: 10.1016/s0360-3016(03)00819-8. PMID 14697445
- [Background] Hingorani M, Colley WP, Dixit S, Beavis AM. Hypofractionated radiotherapy for glioblastoma: strategy for poor-risk patients or hope for the future? Br J Radiol. 2012 Sep;85(1017):e770-81. doi: 10.1259/bjr/83827377. PMID 22919020
- [Background] Laperriere N, Zuraw L, Cairncross G; Cancer Care Ontario Practice Guidelines Initiative Neuro-Oncology Disease Site Group. Radiotherapy for newly diagnosed malignant glioma in adults: a systematic review. Radiother Oncol. 2002 Sep;64(3):259-73. doi: 10.1016/s0167-8140(02)00078-6. PMID 12242114
- [Background] Roa W, Kepka L, Kumar N, Sinaika V, Matiello J, Lomidze D, Hentati D, Guedes de Castro D, Dyttus-Cebulok K, Drodge S, Ghosh S, Jeremic B, Rosenblatt E, Fidarova E. International Atomic Energy Agency Randomized Phase III Study of Radiation Therapy in Elderly and/or Frail Patients With Newly Diagnosed Glioblastoma Multiforme. J Clin Oncol. 2015 Dec 10;33(35):4145-50. doi: 10.1200/JCO.2015.62.6606. Epub 2015 Sep 21. PMID 26392096
- [Background] Roa W, Brasher PM, Bauman G, Anthes M, Bruera E, Chan A, Fisher B, Fulton D, Gulavita S, Hao C, Husain S, Murtha A, Petruk K, Stewart D, Tai P, Urtasun R, Cairncross JG, Forsyth P. Abbreviated course of radiation therapy in older patients with glioblastoma multiforme: a prospective randomized clinical trial. J Clin Oncol. 2004 May 1;22(9):1583-8. doi: 10.1200/JCO.2004.06.082. Epub 2004 Mar 29. PMID 15051755
- [Background] Malmstrom A, Gronberg BH, Marosi C, Stupp R, Frappaz D, Schultz H, Abacioglu U, Tavelin B, Lhermitte B, Hegi ME, Rosell J, Henriksson R; Nordic Clinical Brain Tumour Study Group (NCBTSG). Temozolomide versus standard 6-week radiotherapy versus hypofractionated radiotherapy in patients older than 60 years with glioblastoma: the Nordic randomised, phase 3 trial. Lancet Oncol. 2012 Sep;13(9):916-26. doi: 10.1016/S1470-2045(12)70265-6. Epub 2012 Aug 8. PMID 22877848
- [Background] Keime-Guibert F, Chinot O, Taillandier L, Cartalat-Carel S, Frenay M, Kantor G, Guillamo JS, Jadaud E, Colin P, Bondiau PY, Menei P, Loiseau H, Bernier V, Honnorat J, Barrie M, Mokhtari K, Mazeron JJ, Bissery A, Delattre JY; Association of French-Speaking Neuro-Oncologists. Radiotherapy for glioblastoma in the elderly. N Engl J Med. 2007 Apr 12;356(15):1527-35. doi: 10.1056/NEJMoa065901. PMID 17429084
- [Background] Athanassiou H, Synodinou M, Maragoudakis E, Paraskevaidis M, Verigos C, Misailidou D, Antonadou D, Saris G, Beroukas K, Karageorgis P. Randomized phase II study of temozolomide and radiotherapy compared with radiotherapy alone in newly diagnosed glioblastoma multiforme. J Clin Oncol. 2005 Apr 1;23(10):2372-7. doi: 10.1200/JCO.2005.00.331. PMID 15800329
- [Background] Stupp R, Hegi ME, Mason WP, van den Bent MJ, Taphoorn MJ, Janzer RC, Ludwin SK, Allgeier A, Fisher B, Belanger K, Hau P, Brandes AA, Gijtenbeek J, Marosi C, Vecht CJ, Mokhtari K, Wesseling P, Villa S, Eisenhauer E, Gorlia T, Weller M, Lacombe D, Cairncross JG, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumour and Radiation Oncology Groups; National Cancer Institute of Canada Clinical Trials Group. Effects of radiotherapy with concomitant and adjuvant temozolomide versus radiotherapy alone on survival in glioblastoma in a randomised phase III study: 5-year analysis of the EORTC-NCIC trial. Lancet Oncol. 2009 May;10(5):459-66. doi: 10.1016/S1470-2045(09)70025-7. Epub 2009 Mar 9. PMID 19269895
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Cabrera AR, Kirkpatrick JP, Fiveash JB, Shih HA, Koay EJ, Lutz S, Petit J, Chao ST, Brown PD, Vogelbaum M, Reardon DA, Chakravarti A, Wen PY, Chang E. Radiation therapy for glioblastoma: Executive summary of an American Society for Radiation Oncology Evidence-Based Clinical Practice Guideline. Pract Radiat Oncol. 2016 Jul-Aug;6(4):217-225. doi: 10.1016/j.prro.2016.03.007. Epub 2016 Mar 31. PMID 27211230
- [Background] Central Brain Tumor Registry of the United States (CBTRUS) CBTRUS statistical report: primary brain and central nervous system tumors diagnosed in the United States in 2004-2008. Hinsdale, IL: Central Brain Tumor Registry of the United States; 2012. Feb, pp. 1-58.
- [Background] Wrensch M, Minn Y, Chew T, Bondy M, Berger MS. Epidemiology of primary brain tumors: current concepts and review of the literature. Neuro Oncol. 2002 Oct;4(4):278-99. doi: 10.1093/neuonc/4.4.278. PMID 12356358
- See also: Related Info — https://www.jdyy.cn/